CLINICAL TRIAL: NCT06312228
Title: The Effect of the Helper Skin Tap Technique and Buzzy® Application on the Level of Pain and Anxiety Experienced by Children During Vaccination
Brief Title: The Effect of the Helper Skin Tap Technique and Buzzy® During Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Duygu Sonmez Duzkaya, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/05
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Child, Only
Keywords: pain; fear; Buzzy; Helfer skin tap teknik
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Helper Skin Tap Technique Group (Experimental): Before the vaccine injection, body weight, height and physiological parameters (pulse, blood pressure, SpO2, body temperature) were measured and behavioural pain responses were evaluated by the child, nurse and parent using the Wong-Baker pain scale and fear scale. Slow tapping was performed with rhythmic tapping movements on the left deltoid muscle where the vaccine will be administered to the children. When the needle was to be inserted into the deltoid muscle, the tapping was slightly increased and the needle entry was made with the same movement. After the vaccine injection was given, the needle was rapidly withdrawn from the muscle by increasing the tapping movements while the needle was withdrawn.
  Interventions: Other: Helfer Skin Tap
- Buzzy Group (Experimental): Before the vaccine injection, body weight, height and physiological parameters (pulse, blood pressure, SpO2, body temperature) were measured and behavioural pain responses were evaluated by the child, nurse and parent using the Wong-Baker pain scale and fear scale. The ice pack previously removed from the deep freezer was kept at room temperature for 10 minutes and the hole in the ice pack wing was placed on the hook behind the Buzzy®. The Buzzy® was placed on the left arm deltoid muscle and activated and kept for 30 seconds. After 30 seconds, Buzzy® was pulled up 1 centimetre (cm) and the MMR vaccine injection was administered to the area corresponding to the left deltoid muscle. After the vaccine injection, Buzzy® was pulled to the injection site and kept for another 30 seconds.
  Interventions: Other: Buzzy
- Control Group (No Intervention): Before the vaccine injection, body weight, height and physiological parameters (pulse, blood pressure, SpO2, body temperature) were measured and behavioural pain responses were evaluated by the child, nurse and parent using the Wong-Baker pain scale and fear scale. MMR vaccine injection was routinely administered in the area corresponding to the left deltoid muscle without any intervention or application to the injection site.

INTERVENTIONS:
Other: Helfer Skin Tap — Slow tapping was performed with rhythmic tapping movements on the left deltoid muscle where the vaccine will be administered to the children. When the needle was to be inserted into the deltoid muscle, the tapping was slightly increased and the needle entry was made with the same movement. After the vaccine injection was given, the needle was rapidly withdrawn from the muscle by increasing the tapping movements while the needle was withdrawn.
  Arms: Helper Skin Tap Technique Group
Other: Buzzy — The ice pack previously removed from the deep freezer was kept at room temperature for 10 minutes and the hole in the ice pack wing was placed on the hook behind the Buzzy®. The Buzzy® was placed on the left arm deltoid muscle and activated and kept for 30 seconds. After 30 seconds, Buzzy® was pulled up 1 centimetre (cm) and the MMR vaccine injection was administered to the area corresponding to the left deltoid muscle. After the vaccine injection, Buzzy® was pulled to the injection site and kept for another 30 seconds.
  Arms: Buzzy Group

SUMMARY:
Aim: This randomised controlled experimental study was conducted to determine the effect of Helfer Skin Tap Technique and Buzzy® application on the pain level during measles-mumps-rubella-mumps (MMR) vaccine injection in 4-year-old children.Method: The study was a randomised controlled experimental study. The sample of the study consisted of 96 children (buzzy: 32, helfer skin tap: 32, control: 32) who underwent MMR vaccination at Bakırköy Family Health Centre No. 9 between May 2023 and October 2023. Data Collection Form, Wong-Baker pain scale, Fear scale and Buzzy® device were used as data collection tools. Buzzy® and Helfer skin tap technique were applied to the children in the intervention group before and after the vaccine injection, while routine vaccine injection was applied to the children in the control group. Children's pain and fear responses were evaluated by the nurse and parents before and after vaccine injection, and physiological parameters were evaluated by the nurse before and after vaccine injection.

DETAILED DESCRIPTION:
This randomised controlled experimental study was conducted to determine the effect of Helfer Skin Tap Technique and Buzzy® application on the pain level during measles-mumps-rubella-mumps (MMR) vaccine injection in 4-year-old children.

Materials and Methods Setting The sample of the study consisted of 96 children (buzzy: 32, helfer skin tap: 32, control: 32) who underwent MMR vaccination at Bakırköy Family Health Centre No. 9 between May 2023 and October 2023.

Sample The population of the study, which was planned as a randomised controlled experimental study, consisted of 4-year-old children who applied to Bakırköy Family Health Centre (FHC) No. 9 for MMR vaccination. According to the power analysis for the sample size in line with the literature (Mahato and Thakur 2019; Şıktaş and Uysal 2023), the power of the sample was calculated with the G*Power 3.1 programme. With a Type I error of 0.05 and a test power of 0.80 (α= 0.05, 1-β= 0.80), the minimum sample size (30 children in each group) was calculated as 90 children. Considering the losses that may occur from the sample for any reason during the study period, the study was completed with 96 children, including 32 children in the study and control groups.

Data Collection In the study, children who came to the Family Health Centre for MMR vaccination were first evaluated in terms of sampling criteria, and infants who did not meet the criteria were excluded from the study. The nurses who collected and administered the data are different. According to the childhood vaccination calendar of the Ministry of Health, MMR, quadrivalent mixed vaccine (DaBT-IPA (diphtheria, acellular pertussis, tetanus, inactive polio) are administered at the age of 4 years. The infants included in the study were first given MMR vaccine in the left arm and the other vaccine was given in the leg 10 minutes after the end of the administration.

Application MMR vaccine was administered according to the vaccine administration technique in the Ministry of Health's Expanded Immunisation Programme (2009) Circular. Vaccines are stored in the refrigerator under cold chain conditions between +2 0C - +8 0C. Before vaccine injection, it was ensured that the vaccination room was well lit and warm, and children were in a comfortable environment. The children in the Helfer Skin Tap Technique, buzzy and control group, who met the sampling criteria, were first examined by the family physician, and the parents of the children who did not have any objection to vaccination were informed about the research and their verbal and written consent was obtained and then the data collection form was filled out. Before the vaccine injection, body weight, height and physiological parameters (pulse, blood pressure, SpO2, body temperature) were measured and behavioural pain responses were evaluated by the child, nurse and parent using the Wong-Baker pain scale and fear scale. The child was first seated on the parent's lap (on the knee) and the holding position was adjusted. The child's legs were placed between the parent's legs and the arms were wrapped around the parent to hold the child. After the vaccine injection, pain and fear responses were evaluated by the nurse and parent using the Wong-Baker pain scale and fear scale. In addition, physiological parameters of the children were also measured and recorded.

STATISTICAL ANALYSIS Statistical analyses were performed using R vers. 2.15.3 program Minimum, maximum, mean, standard deviation, median, first quartile, third quartile, frequency, and percentage were used to report the study data. The Shapiro-Wilk test and graphical analysis were used to evaluate the compliance of quantitative data with normal distribution. A dependent groups t-test was used to compare the values before and after the intervention. An independent groups t-test was used to evaluate normally distributed variables between two groups. One-way analysis of variance was used in the evaluations of variables with normal distribution between more than two groups. The Mann-Whitney U test evaluated variables that did not show normal distribution between the two groups. The Kruskal-Wallis test was used in the evaluations of variables that did not show normal distribution between more than two groups. Pearson correlation analysis was used to determine the relationship between quantitative variables. The Pearson chi-square test, Fisher-Freeman-Halton exact test, and Fisher's exact test were used to compare qualitative variables. Statistical significance was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* The child being at least 4 years old,
* The administration of the DTP vaccine,

  * Being at an appropriate weight for their age,
  * The child not having received any analgesic medication during the day,
  * The willingness of the parent to participate in the research

Exclusion Criteria:

- Having a neurological illness,

* Having a chronic illness,
* Having an allergy (egg allergy),
* Having a body temperature above 37.5 degrees Celsius

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Child Information Form | 1 day
  The information form has been prepared by reviewing the literature on the subject (Canbulat and Bal 2015; Canbulat et al 2014) and includes the child's age, gender, height, weight, presence of other children in the family, physiological parameters before and after vaccination injection, Wong-Baker pain score, and Fear score evaluated by the nurse, parent, and child before and after the vaccination injection. There are a total of 5 questions in the data collection form.
Wong-Baker Scale (Pain Facial Expression Scale) | 1 day
  The Wong-Baker scale consists of faces representing increasing levels of pain from zero to five, moving from left to right. The face on the far left has a smiling expression, indicating a pain-free condition, while the face on the far right has a crying expression, representing the most severe pain. Each facial expression is accompanied by a brief description explaining the pain intensity: 0 - no pain, 1 - mild pain, 2 - a bit more pain, 3 - even more pain, 4 - quite a lot of pain, 5 - the most severe pain.
Child Fear Scale | 1 day
  The Child Fear Scale is used to assess the anxiety levels of children with five face shapes scored between 0-4: 0 = no anxiety, and 4 = severe anxiety. The scale can be evaluated by both the child and the researcher before, during, and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Background] Therese, A. M., & Devi, S. (2014). Effectiveness of Helfer skin tap technique and routine technique on pain reduction among patients receiving intramuscular injection at Government General Hospital, Puducherry. Int J Sci Res, 3(10).
- [Background] Jose, R. M., Sulochana, B., & Shetty, S. (2012). Effectiveness of Skin Tap Technique in Reducing Pain Response. International Journal of Nursing Education, 4(1).
- [Background] Mahato, E. (2019). Effectiveness of Helfer's Skin Tap Technique Versus Routine Technique on Pain Reduction among Patient's Receiving Intramuscular Injections. International Journal of Nursing Education, 11(1),41-44.
- [Background] Taddio A, McMurtry CM, Shah V, Riddell RP, Chambers CT, Noel M, MacDonald NE, Rogers J, Bucci LM, Mousmanis P, Lang E, Halperin SA, Bowles S, Halpert C, Ipp M, Asmundson GJG, Rieder MJ, Robson K, Uleryk E, Antony MM, Dubey V, Hanrahan A, Lockett D, Scott J, Bleeker EV; HELPinKids&Adults. Reducing pain during vaccine injections: clinical practice guideline. CMAJ. 2015 Sep 22;187(13):975-982. doi: 10.1503/cmaj.150391. Epub 2015 Aug 24. No abstract available. PMID 26303247
- [Background] Shah V, Taddio A, McMurtry CM, Halperin SA, Noel M, Pillai Riddell R, Chambers CT; HELPinKIDS Team. Pharmacological and Combined Interventions to Reduce Vaccine Injection Pain in Children and Adults: Systematic Review and Meta-Analysis. Clin J Pain. 2015 Oct;31(10 Suppl):S38-63. doi: 10.1097/AJP.0000000000000281. PMID 26201016
- [Background] Noel M, Chambers CT, McGrath PJ, Klein RM, Stewart SH. The influence of children's pain memories on subsequent pain experience. Pain. 2012 Aug;153(8):1563-1572. doi: 10.1016/j.pain.2012.02.020. Epub 2012 May 3. PMID 22560288
- [Background] Koc T, Gozen D. The Effect of Foot Reflexology on Acute Pain in Infants: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2015 Oct;12(5):289-96. doi: 10.1111/wvn.12099. Epub 2015 Jul 28. PMID 26220257